CLINICAL TRIAL: NCT05968118
Title: A Double-Blind, Randomized, Placebo-Controlled, Single Center Study to Assess the Angiogenesis and Blood Perfusion Effect of NL003 in Patients With Critical Limb Ischemia by PETCT-RGD and MIBI
Brief Title: Angiogenesis and Blood Perfusion Effect of HGF Gene Therapy in PAD Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL003-PAD-III-3
Record Dates: First submitted 2023-01-04; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; Hepatocyte Growth Factor; NL003; Gene therapy; PET/CT-RGD; MIBI
MeSH Terms: conditions — Peripheral Arterial Disease; Deafness, Autosomal Recessive 39 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational product (Experimental): Patients in this treatment group will receive 8mg NL003 respective in D0、14、28
  Interventions: Drug: NL003
- Placebo (Placebo Comparator): Patients in this group will receive normal saline respective in D0、14、28
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NL003 — Day 0: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 14: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 28: 8mg of NL003 (32 injections of 0.5ml of NL003)
  Other Names: HGF plasmid; pCK-HGF-X7
  Arms: investigational product
Drug: Placebo — Day 0: 16ml of Normal Saline (32 injections ) Day 14: 16ml of Normal Saline (32 injections ) Day 28: 16ml of Normal Saline (32 injections ) Other Name: Placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether PET/CT-RGD or MIBI can be used for the angiogenesis assessment of NL003 in PAD patients.

DETAILED DESCRIPTION:
Hepatocyte growth factor (HGF) gene therapy has been shown to be a potential choice for CLI patients without surgical option. NL003, which is a DNA plasmid that contains novel genomic cDNA hybrid human HGF coding sequence (HGF-X7) expressing two isoforms of HGF, HGF 728 and HGF 723. Animal studies showed that NL003 inducing angiogenesis in the affected limb and result in an increase in tissue perfusion. Our previous phase II clinical trial has suggested the successful limb-salvaging capacity of NL003 in treatment of patients with CLTI.

In this study we will use 68Ga RGD PET/CT and 99mTc MIBI SPECT imaging methods to evaluate the effect of NL003 on angiogenesis and lower limb blood flow perfusion during the treatment of chronic lower limb ischemia, and evaluated the effectiveness and safety of the drug. The subjects will be randomly divided into the investigational drug group and the placebo group in a 1:1 ratio. NL003 or placebo will be injected into the muscle of the affected limb on D0, D14 and D28, 0.5mg/0.5mL/site, total 8mg, 32 sites. PET/CT will be measured on D14, D42 before drug administration, MIBI SPECT imaging will be collected on D60.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years, diagnosed with chronic lower limb ischemia;
2. According to DSA or CTA，severe stenosis (≥70%) or occlusion of one or more branches of superficial femoral artery, popliteal artery, anterior tibial artery, posterior tibial artery, and peroneal artery.
3. Patients with obvious symptoms of lower limb ischemia, including severe claudication, resting pain, ulcers, or gangrene.
4. Agree to use appropriate contraceptive methods during the trial; Female subjects of reproductive age, blood pregnancy test negative.
5. Signing the informed consent.
6. Can complete PETCT-RGD check and MIBI check;

Exclusion Criteria:

1. The foot or lower limb infection cannot be controlled, and amputation may be accepted within 3 months.
2. Those with cerebral infarction, cerebral hemorrhage, heart failure, unstable angina, acute myocardial infarction, and serious arrhythmia within 3 months;
3. Tumor patients diagnosed with malignant tumor or suspected of having malignant tumor after tumor screening;
4. Main iliac artery stenosis ≥ 70%;
5. Refractory hypertension (taking three or more antihypertensive drugs, systolic blood pressure ≥ 180mmHg or diastolic blood pressure ≥ 110mmHg);
6. Anti HIV antibody positive person, anti hepatitis C antibody positive person and RNA positive person, hepatitis B surface antigen positive person (if the subject is HBsAg positive, and judging by peripheral blood HBV DNA, the researcher believes that the subject is in a stable period of chronic hepatitis B, which will not increase the risk of the subject, the subject can be selected)
7. Patients with poor blood glucose control after treatment (HbA1c>10%);
8. Persons allergic to contrast medium
9. The investigator believes that the patient's complications affect the evaluation of safety and effectiveness, or the expected survival period is less than 12 months;
10. Those who regularly drink more than 14 units of alcohol (1 unit=360 mL beer or 45 mL liquor or 150 mL wine with 40% alcohol) or drug abusers within 12 months before signing the informed consent form;
11. Acute lower limb ischemia or acute aggravation of chronic lower limb ischemia;
12. Those who received vascular reconstruction of the affected limb within 4 weeks before the informed consent form and whose blood supply improved after the operation
13. Serious liver or kidney disease or severe anemia judged by the investigator;
14. Those who cannot correctly describe symptoms and emotions;
15. Those who participated in other clinical trials within 3 months before signing the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes of the new blood vessels number | Day 14、Day 42
  changes in the number of new blood vessels measured by PETCT-RGD on D14 and D42, compare with that of the baseline.
Changes of local blood perfusion | Day 60
  the changes of local blood perfusion measured by MIBI on D60, compare with that of baseline.

SECONDARY OUTCOMES:
Changes to the ABI from the baseline | Day 60
  Ankle-brachial index (ABI) refers to the ratio of systolic blood pressure of the anterior tibial artery (dorsal foot artery) or posterior tibial artery to the systolic blood pressure of the brachial artery.Participants were tested for ankle-brachial index (ABI).
Laser Speckle Imaging changes in blood flow from the baseline | Day 60
  Laser Speckle Imaging changes in blood flow from the baseline was measured on D60.
Changes of pain score from the baseline | Day 14、Day 28、Day 42、Day 60、Day 90
  The severity of critical Limb ischemia was assessed by Rutherford grading at screening、D14、D28、D42、D60、D90
Gangrene /Ulcer changes from the baseline | Day 14、Day 28、Day 42、Day 60、Day 90
  Changes in the area of ulcer or gangrene from baseline after use of the study drug
Changes in quality of life scores from baseline | Day 60
  The quality of life score questionnaire was conducted to evaluate the subjective perception of Critical Limb Ischemia, including the subjects' perception of quality of life, health, or other aspects of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No